CLINICAL TRIAL: NCT04003025
Title: Body Composition Evaluation as a Prognosis Determinant in Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Body Composition and Prognosis in Head and Neck Squamous Cell Carcinoma (HNSCC)
Acronym: HNCAX01
Status: Withdrawn | Type: Observational
Why Stopped: The proposed analysis was not feasible.
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: NP 1454/19
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study in patients with cancer of the oral cavity, pharynx, and larynx. Imaging exams of these patients will be analyzed with the objective of developing and validating a clinically applicable method for evaluation of cachexia and/or sarcopenia in a patient with head and neck cancer from musculature imaging of the neck. Indeed, the prognostic influence of body composition will be evaluated.

DETAILED DESCRIPTION:
Epidermoid carcinoma (SCC) is the predominant histology of cancers of the oral cavity, pharynx, and larynx. In Brazil, 11,200 new cases of oral cavity cancer are estimated in men and 3,500 in women for each year of the 2018-2019 biennium. The disease causes high mortality and morbidity, affecting swallowing and dysphagia, leading to weight loss and cachexia. Cancer cachexia is marked by involuntary muscle loss leading to progressive functional impairment and can not be reversed by traditional nutritional support. Recent publications show that muscle mass can predict certain outcomes such as survival. Methods for assessing body composition have been developed and validated for research, and the area of a skeletal muscle, which can be measured by cross-sectional images, is a valid marker of total body mass. The CT evaluation of the region of the third and fourth lumbar vertebra (L3-L4) are accurate and accepted as a method for evaluating body composition. However, given the locoregional nature of the dissemination of this SCC, usually the L3-L4 level is not available on CT, and this is a limitation for the use of CT to assess cachexia in these patients. This study will be divided into three steps. In the first step, 20 patients with cross-sectional CT images of patients with head and neck cancer diagnosis will be selected to verify the intra-class variation at different evaluation times. The second step aims to evaluate the correlation of the muscular area obtained through the L3 region with the area of the neck muscles. The third step will evaluate the prognostic role of the neck muscle area of HNSCC patients. The area of the neck muscle of the first CT scan obtained prior to the beginning of treatment will be evaluated and the ratio of this area with the survival rate will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have histological or cytological evidence of oropharynx squamous cell carcinoma, oral cavity, larynx or hypopharynx, locally advanced treated only at Sao Paulo Cancer Institute (ICESP).

Exclusion Criteria:

* patients with no tomography available.
* head and neck cancer with tumor at other sites such as thyroid, paranasal sinus, skin and nasopharynx, or other histology other than squamous cell carcinoma

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have histological or cytological evidence of oropharynx squamous cell carcinoma, oral cavity, larynx or hypopharynx, locally advanced treated only at Sao Paulo Cancer Institute (ICESP).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival in HNSCC | 1 year
  Survival will be measured to understand the prognostic impact of skeletal muscle index in HNSCC

SECONDARY OUTCOMES:
Skeletal muscle index of L3 and C3 | 1 years
  The correlation of L3 and C3 will measured as alternative areas of skeletal muscle index to evaluate sarcopenia/cachexia.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo, Brazil